CLINICAL TRIAL: NCT02414607
Title: Effect of Elderberry Juice on Cognition and Inflammation in Patients With Mild Cognitive Impairment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, David Beversdorf, Associate Professor: Radiology, Neurology, Psychology, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1211953
Record Dates: First submitted 2015-03-20; First posted 2015-04-13 (Estimated); Results first posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-05

CONDITIONS: Mild Cognitive Impairment
Keywords: Elderberry juice; Alzheimer's; Inflammation
MeSH Terms: conditions — Cognitive Dysfunction; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elderberry Juice (Experimental): Participants will drink 5ml of elderberry juice, diluted in 8oz of water, 3 times per day for three months.
  Interventions: Biological: Elderberry Juice
- Placebo (Placebo Comparator): Participants will drink 5ml of colored water, diluted in 8oz of water, 3 times per day for three months.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Elderberry Juice
  Arms: Elderberry Juice
Other: Placebo
  Arms: Placebo

SUMMARY:
Elderberries (Sambuci fructus) have been shown in a number of studies to have significant anti-inflammatory and antioxidant effects. Multiple human and animal studies have supported the anti-inflammatory and antioxidant effects of elderberry preparations and it has been used in natural medicine for hundreds of years. Studies examining factors that may decrease the risk of Alzheimer's disease have revealed that drinking juices with similar properties to elderberries is one of the most reliable way to decrease risk. As such the investigators wish to determine the effects of elderberry juice on cognitive decline in a group of subjects at high risk for Alzheimer's disease, those with mild cognitive impairment. Elderberry juice is a commercially available nutritional supplement and easily available to this population.

ELIGIBILITY:
Inclusion Criteria:

* CDR score of 0.5
* MMSE of at least 24
* Age 50 or older

Exclusion Criteria:

* Known history of sensitivity to elderberry products.
* Diabetes.
* Bleeding disorder.
* Current Pregnancy.
* Known allergy to honeysuckle.
* Currently making changes to other drugs that might affect cognitive performance (subjects showing the greatest cognitive decline and other signs of Alzheimer's disease may be prescribed cholinesterase inhibitors as this is a standard of care for Alzheimer's disease but not MCI).
* Presence of any condition the health professional believes will impair ability to complete study procedures (ex. terminal illness, comorbid major psychiatric disorders such as schizophrenia, or drug abuse).
* Potentially confounding neurodegenerative diseases (e.g. MS).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-09; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Q Beversdorf, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Hospital, Columbia, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Elderberry Juice: Participants will drink 5ml of elderberry juice, diluted in 8oz of water, 3 times per day for three months.
  Elderberry Juice
- Placebo: Participants will drink 5ml of colored water, diluted in 8oz of water, 3 times per day for three months.
  Placebo
Period: Overall Study
Arm/Group | Elderberry Juice | Placebo
Started | 11 | 13
Completed | 9 | 11
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elderberry Juice | Placebo | Total
Number analyzed (Participants) | 11 | 13 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 10 | 13 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.45 (8.47) | 76.23 (7.73) | 76.33 (6.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 3 | 7 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 13 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 13 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 13 | 24

OUTCOME MEASURES:

1. Primary Outcome: Visuospatial Problem Solving Battery (VSP)
Description: Problem solving task for detecting non-memory impairments in MCI. Change in score is the outcome measure. The task is a timed task, with the outcome measured in seconds. Each item was allowed 240 seconds for solution, with times averaged for items. Therefore, there was a range of 0-240 with lower being better.
Time Frame: 12 wks, 6 mos
Measure: Mean (Standard Error); unit: Mean Difference Score (VPS Total Score)
Arm/Group | Elderberry Juice | Placebo
Number analyzed (Participants) | 11 | 13
Mean Difference Score (VPS Total Score)
  12 week change from baseline | .30 (.52) | .29 (.47)
  6 month change from baseline | .097 (.44) | .52 (.38)

2. Secondary Outcome: Clinical Dementia Rating (CDR) Scale
Description: Assesses memory, orientation, judgement and problem solving, community affairs, home/hobbies, personal care. Change in CDR was the outcome. CDR ranges from 0 to 3, with 3 being worse.
Time Frame: 12 wks, 6 mos
Measure: Mean (Standard Error); unit: Mean difference on CDR scale
Arm/Group | Elderberry Juice | Placebo
Number analyzed (Participants) | 11 | 13
Mean difference on CDR scale
  Change from Baseline at 12 weeks | 0 (0) | 0 (0)
  Change from Baseline at 6 months | 0 (0) | 0 (0)

3. Secondary Outcome: Mini-Mental State Examination (MMSE)
Description: Screening for cognitive impairment sampling functions including arithmetic, memory and orientation. Change in MMSE was the outcome. the MMSE is a scale from 0 to 30 with a higher score being better.
Time Frame: 12 wks, 6 mos
Measure: Mean (Standard Error); unit: Mean Difference Score (MMSE)
Arm/Group | Elderberry Juice | Placebo
Number analyzed (Participants) | 11 | 13
Mean Difference Score (MMSE)
  Change from baseline at 12 weeks | .03 (.73) | .29 (.66)
  Change from baseline at 6 months | -1.01 (.90) | .06 (.82)

4. Secondary Outcome: Hopkins Verbal Learning Test (HVLT)
Description: Assesses verbal learning and memory. Change in the HVLT was the outcome measure. The range for the HVLT is 0-36 with higher representing better memory.
Time Frame: 12 wks, 6 mos
Measure: Mean (Standard Error); unit: Mean Difference Score (HVL Free Recall)
Arm/Group | Elderberry Juice | Placebo
Number analyzed (Participants) | 11 | 13
Mean Difference Score (HVL Free Recall)
  Change from baseline at 12 weeks | -.50 (.43) | .46 (.40)
  Change from baseline at 6 months | -19 (.33) | .27 (.29)

5. Secondary Outcome: Boston Naming Test (BNT)
Description: Measures word retrieval. Change in the BNT is the primary outcome measure. The range is 0-60 with higher representing better performance.
Time Frame: 12 wks, 6 mos
Measure: Mean (Standard Error); unit: Mean Difference Score (BNT Total)
Arm/Group | Elderberry Juice | Placebo
Number analyzed (Participants) | 11 | 13
Mean Difference Score (BNT Total)
  Change from baseline at 12 weeks | 1.38 (.65) | .94 (.59)
  Change from baseline at 6 months | .96 (.54) | 1.60 (.49)

6. Secondary Outcome: Rey Complex Figure Task (Rey)
Description: Participants reproduce complicated line drawings. Change in the Rey was the primary outcome measure. The range of the Rey is 0-36 with a higher score being better performance.
Time Frame: 12 wks, 6 mos
Measure: Mean (Standard Error); unit: Mean Difference Score (REY Copy Score)
Arm/Group | Elderberry Juice | Placebo
Number analyzed (Participants) | 11 | 12
Mean Difference Score (REY Copy Score)
  Change from baseline at 12 weeks | -1.03 (1.43) | 1.41 (1.35)
  Change from baseline at 6 months | -.54 (1.61) | -1.72 (.27)

7. Secondary Outcome: Anagrams
Description: Rearranging letters to form words. Change in performance is the primary outcome measure. The task is timed, with each anagram allowed 120 seconds, so each word has a range of 0-120 seconds, and the average for the latency was calculated, for a range of 0-120 with lower numbers being better.
Time Frame: 12 wks, 6 mos
Measure: Mean (Standard Error); unit: Mean Difference Score (Anagrams Total)
Arm/Group | Elderberry Juice | Placebo
Number analyzed (Participants) | 11 | 12
Mean Difference Score (Anagrams Total)
  Change from baseline at 12 weeks | -1.81 (.13) | 2.70 (.99)
  Change from baseline at 6 months | -.41 (.95) | 1.67 (.86)

8. Secondary Outcome: Instrumental Activities of Daily Living Scale (IADLS)
Description: Assesses daily self-care activities. Change in the IADLS is the primary outcome. Total items were added together for this use of the task, so the range was from 0 to 23, with higher being better.
Time Frame: 12 wks, 6 mos
Measure: Mean (Standard Error); unit: Mean Difference Score (IADL)
Arm/Group | Elderberry Juice | Placebo
Number analyzed (Participants) | 11 | 12
Mean Difference Score (IADL)
  Change from baseline at 12 weeks | .40 (.69) | -.34 (.59)
  Change from baseline at 6 months | -30 (.66) | -44 (.60)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Serious adverse events or adverse events were documented.
Arm/Group | Elderberry Juice | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/13
Other Adverse Events (participants affected / at risk) | 0/11 | 1/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elderberry Juice (N=11) | Placebo (N=13)
Non-serious adverse event (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Acute skin rash

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-05-11): https://cdn.clinicaltrials.gov/large-docs/07/NCT02414607/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/07/NCT02414607/SAP_001.pdf